CLINICAL TRIAL: NCT03512912
Title: Transcutaneous Electrostimulation of the Calf Muscle and Supervised Walking Therapy for Intermittent cLAudication
Brief Title: Transcutaneous Electrostimulation for Intermittent Claudication Supervised Walking Therapy for Intermittent cLAudication
Acronym: TESLA
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Heinrich-Heine University, Duesseldorf (Other)
Responsible Party: Principal Investigator, Dr. Philip Düppers, Dr. med., Heinrich-Heine University, Duesseldorf
Other Study IDs: TESLA
Record Dates: First submitted 2018-04-19; First posted 2018-05-01 (Actual); Last update posted 2018-05-07 (Actual); Status verified 2018-05

CONDITIONS: Intermittent Claudication; Peripheral Arterial Disease
MeSH Terms: conditions — Intermittent Claudication; Peripheral Arterial Disease

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

INTERVENTIONS:
Device: transcutaneous electrical calf muscle stimulation + supervised walking therapy — transcutaneous electrical calf muscle stimulation + supervised walking therapy

SUMMARY:
Prospective mono-centric trial on patients with peripheral arterial disease and intermittent claudication that receive supervised exercise therapy (group 1) vs. supervised exercise therapy + daily transcutaneous electro-stimulation of the calf muscles.

DETAILED DESCRIPTION:
The investigators conduct a prospective mono-centric trial on all patient with peripheral arterial disease with intermittent claudication that receive supervised exercise therapy (SET) and additional transcutaneous electric stimulation (TES) of the calf muscle. SET program consists in once weekly walking training for 75 min under supervision of a professional trainer. Patients are encouraged to continue the training modules at home. TES is performed using the mobile "Veinoplus arterial" device (AdRem Technology, France) on a daily base for 60-120 min at home. Patient outcome will be compared to the retrospectively analyzed results of patients, that received the same SET program alone in the past.

ELIGIBILITY:
Inclusion Criteria:

* intermittent claudication due to peripheral arterial disease
* ankle brachial index </=0.9
* occlusion or stenosis of the superficial femoral artery

Exclusion Criteria:

* rest pain or peripheral arterial lesions
* contraindications for supervised walking therapy
* non-vascular conditions that limit patients´ walking ability
* patients that have already received supervised walking therapy
* occlusion of the deep femoral artery
* occlusion or high-grade stenoses of the iliac arteries
* stroke in the last 12 months
* premenopausal women
* diabetes mellitus, dialysis, sclerodermia and other conditions that impair leg perfusion
* active cilostazol therapy or alprostadil-infusion in the last 3 months
* pacemaker, defibrillator systems, life vest
* visible muscle contraction is not achieved without pain

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All patients of our department of vascular end endovascular surgery, university hospital Dusseldorf with the above mentioned inclusion criteria.
Sampling Method: Non-Probability Sample
Enrollment: 20 (Estimated)
Dates: Start 2018-05 (Estimated); Primary Completion 2020-05 (Estimated); Study Completion 2020-05 (Estimated)

PRIMARY OUTCOMES:
Walking distance | 6 months
  Measurement of the pain-free and absolute walking distance on a standardized constant load treadmill test

CONTACTS AND LOCATIONS:
Overall Officials: Philip Düppers, MD, Principal Investigator — Department of Vascular and Endovascular Surgery
Locations (1):
- University Hospital Dusseldorf, Department of Vascular and Endovascular Surgery, Düsseldorf, North Rhine-Westphalia, Germany

IPD SHARING:
Plan to Share IPD: No